CLINICAL TRIAL: NCT05125562
Title: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles Infusion Treatment for Mild-to-Moderate COVID-19: A Phase II Clinical Trial
Brief Title: Extracellular Vesicles Infusion Treatment for Mild-to-Moderate COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor has withdrawn/closed the IND with the FDA. A letter dated 21NOV2022 was submitted to the FDA.
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DB-EF-EMOTECOVID-0006
Expanded Access: NCT04657458 (No longer available)
Record Dates: First submitted 2021-11-11; First posted 2021-11-18 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: ExoFlo; COVID-19; Extracellular Vesicle; Mild
MeSH Terms: conditions — COVID-19; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 100ml normal saline
  Interventions: Drug: ExoFlo
- 10ml ExoFlo (Experimental): 10ml ExoFlo + 90ml normal saline
  Interventions: Drug: ExoFlo
- 15ml ExoFlo (Experimental): 15ml ExoFlo + 85ml normal saline
  Interventions: Drug: ExoFlo

INTERVENTIONS:
Drug: ExoFlo — Patients will be randomized to one of three infusions: (1) Normal Saline 100 mL, (2) Normal saline 90 mL and ExoFlo 10 mL, which is 7x1011 EVs, and (3) Normal saline 85 mL and ExoFlo 15 mL, which is 10.5x1011 EVs. The study intervention will only be dosed on day=1

SUMMARY:
Early Mild Outpatient infusion Therapy with ExoFloTM for COVID-19 (EMOTE COVID-19)

To evaluate the safety and efficacy of intravenous (IV) administration of bone marrow mesenchymal stem cell derived extracellular vesicles, ExoFlo, as treatment for mild-moderate COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for study enrollment includes meeting all the following criteria:

Provision of signed and dated informed consent form (either by the individual or by the individual's healthcare proxy).

Stated willingness to comply with all study procedures and availability for the duration of the study.

Male or female aged 18-85.

COVID-19 positive as defined by positive Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) SARS-CoV-2 determination < 3 days prior to Day of Randomization.

Must have mild or moderate COVID-19 as consistent with NIH definition:

Mild COVID-19: Individuals who have any of the various signs and symptoms of COVID-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and smell) but who do not have shortness of breath, dyspnea, or abnormal chest imaging.

Moderate COVID-19: Individuals who show evidence of lower respiratory disease during clinical assessment or imaging and who have an oxygen saturation (SpO2) ≥94% on room air at sea level.

Duration of illness from acute COVID-19 symptom onset must be 10 days or less.

Only subjects who are not at high risk for progression to severe COVID-19 will be included in the study. See Exclusion Criterion #6.

Subjects who received COVID-19 vaccination are eligible for the study if it is more than 28 days since the last dose of vaccination. COVID-19 vaccination is not necessary for inclusion.

All subjects will need be on < 5 L O2/min to be included or on no oxygen to be enrolled in this study.

If the candidate is either male or female of reproductive potential, he or she must agree to use of double barrier method of highly effective birth control contraception such as condoms with oral contraceptive pill or choose to remain abstinent if already practicing abstinence during the screening period. The duration of required usage of double barrier method OR maintenance of abstinence must include the time from the beginning of the screening period until 90 days following the last dose of the study treatment.

Exclusion Criteria:

* Exclusion from study enrollment includes meeting one or more of the following criteria:

Vulnerable populations such as pregnant patients, children, individuals with severe physical or mental disabilities who cannot provide meaningful consent.

SpO2 < 94% on ambient air.

Active malignancy requiring treatment within the last five years.

Major surgery or physical trauma in the last 3 months, including motor vehicle accidents, assaults, mechanical falls with sequelae of significant bleeding or craniofacial bruising, and surgeries.

All subjects with any comorbidities that may be associated with risk of progression to severe COVID-19 including but not limited to renal dysfunction, hepatic disease, substance abuse, fibromyalgia, heart failure, uncontrolled arrhythmias, any level of dementia, depression, connective tissue diseases, major neuromuscular deficits, and endocrine disorders.

Subjects found to be at high risk for progression to severe COVID-19 will be excluded from the study. These subjects will be referred to outpatient internal medicine clinic for SARS-CoV-2 monoclonal antibody treatment. As defined by the CDC and NIH, high risk for progression to severe COVID-19 is defined by meeting at least one of the following criteria:

Body mass index (BMI) >35

Have chronic kidney disease

Have diabetes

Have immunosuppressive disease

Are currently receiving immunosuppressive treatment

Are >65 years of age

Are >55 years of age AND have

Cardiovascular disease, OR

Hypertension, OR

Chronic obstructive pulmonary disease/other chronic respiratory disease.

Patients who received SARS-CoV-2 monoclonal antibody treatment will be excluded from the study.

Vital sign abnormalities: temperature ≥ 38 °C, temperature < 35 °C; systolic blood pressure (SBP) < 90 mmHg, SBP ≥ 170 mmHg; diastolic blood pressure (DBP) < 50 mmHg, DBP ≥ 100 mmHg; heart rate (HR) < 50 beats per minute (BPM), HR ≥ 120 BPM.

Lab abnormalities: WBC ≥ 12,000 /μL, Creatinine ≥ 1.5 mg/dL, AST ≥ 100 IU/l, and/or ALT ≥ 100 IU/I

Patients who received COVID-19 vaccination within last 28 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-07 (Estimated); Primary Completion 2023-03-07 (Estimated); Study Completion 2023-03-07 (Estimated)

PRIMARY OUTCOMES:
Change in SARS-CoV-2 log viral load from baseline to Day=7 | 61 days
  Change in SARS-CoV-2 log viral load from baseline to Day=7

SECONDARY OUTCOMES:
Change in viral load area under the curve (AUC) from baseline to Day=29 | 61 days
  Change in viral load area under the curve (AUC) from baseline to Day=29
Proportion of patients showing symptom improvement or resolution Day=7, 11, 15 | 61 days
  Proportion of patients showing symptom improvement or resolution Day=7, 11, 15
- Proportion of patients who required COVID-19 related hospitalization or Emergency Department Visit by Day 29 | 61 Days
  - Proportion of patients who required COVID-19 related hospitalization or Emergency Department Visit by Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC

IPD SHARING:
Plan to Share IPD: No